CLINICAL TRIAL: NCT03357328
Title: Therapy Light Rooms for Nursing Home Patients With Dementia - Designing Diurnal Conditions for Improved Sleep, Mood and Behavioural Problems (DEM.LIGHT)
Brief Title: Therapy Light Rooms for Improved Sleep in Dementia Patients
Acronym: DEMLIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBergenDEM.LIGHT; 2016/2246 (Other: Regional committees for medical and health research ethics)
Record Dates: First submitted 2017-11-14; First posted 2017-11-29 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Sleep Fragmentation; Behavioural and Psychiatric Symptoms of Dementia; Dementia
Keywords: Phototherapy; Nursing home; Light therapy
MeSH Terms: conditions — Sleep Deprivation; Dementia

STUDY DESIGN:
Intervention Model Description: 4 nursing home units will receive the intervention (ceiling mounted LED-light in the living room) and 4 will receive the control condition ("standard light"). The trial lasts for 24 weeks. Data will be collected at baseline and after 8, 16 and 24 weeks.
Who Masked: Participant, Care Provider
Masking Description: Although the placebo effect might not be an issue in those with severe dementia, the treatment may affect staff, creating bias such as the Hawthorne effect. Potential changes in staff routines and behaviours in response to the treatment may affect outcome, making a control condition necessary. In this controlled trial, we will compare patients receiving the intervention (therapy light rooms) with control units receiving placebo light ("standard light"). The researchers will install the same standard light solution (100 lux at eye level, 3000K) in all control units. This represents the placebo light intervention, which at the same time ensures a constant standard light condition in all control units.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy light room (Active Comparator): This group (4 NH units, about 35 patients) will receive light therapy administered via LED technology. The light will vary in intensity and colour temperature throughout the day. Ceiling-mounted LED-lights are installed in the living rooms of participating nursing home units. Between 07:00 and 10:00 light of 400 lux at eye level, with 4000 K, will be provided. Between 10:00 and 15:00 the light will comprise 1000 lux at eye level, with 6000 K. From 15:00 to 18:00 the light will comprise 400 lux at eye level and 4000 K. When light is on from 18:00 to 07:00, standard light (about 100 lux at eye level, 3000K) will be administered.
  Interventions: Other: Therapy light room
- Standard light (Placebo Comparator): This group (4 NH units, about 35 patients) will receive "standard light" (100 lux at eye level, 3000K). The light will be administered between 07:00 and 18:00; and the same when light is on between 18:00 to 07:00. This represents the placebo light intervention, which at the same time ensures a constant standard light condition in all control units.
  Interventions: Other: Standard light

INTERVENTIONS:
Other: Therapy light room — See group description
  Arms: Therapy light room
Other: Standard light — See group description
  Arms: Standard light

SUMMARY:
This intervention study will investigate the effect of therapy light rooms on sleep, circadian rhythms, mood, behavioural problems and function in nursing home (NH) patients with dementia.

DETAILED DESCRIPTION:
People with dementia often have fragmented night-time sleep, prolonged night-time awakenings and increased daytime sleep. Behavioural and psychological symptoms of dementia (BPSD) (e.g. agitation, depression) are also common. Noticeably, both sleep problems and BPSD are related to a disturbed circadian rhythm. Light is the most important input to the circadian system, and exposure to sufficient daylight is important for entrainment of the circadian rhythm to the surroundings. Dementia patients living in nursing homes (NH) are less exposed to daylight than dementia patients living at home. Bright light therapy is a promising treatment in these patients as it may improve sleep, BPSD, and independent functioning. However, traditional bright light treatment has not been routinely employed in NH patients or patients with dementia. This may be related to difficulties in achieving adherence to the traditional treatment and thus the benefit of bright light therapy for people with dementia still remains unclear.

DEM.LIGHT uses modern LED (light-emitting diodes) technology that enables light therapy with the least possible interference of the day-to-day life in NHs, as the treatment is not confined to a light source presupposing behavioural compliance. Ceiling-mounted LED-sources can be programmed in terms of timing, light intensity and colour temperature. DEM.LIGHT uses this to provide therapy light rooms with a dynamic light condition that better emulates natural light throughout the day. The study is a cluster-randomized trial evaluating the effect of therapy light rooms on various measures of physical and mental health in NH patients with dementia. Data will be collected at baseline, after 8 and 16 weeks of treatment, and at the end of the intervention period (24 weeks).

ELIGIBILITY:
Inclusion Criteria:

* 60 years or more of age and in long term care (longer than 4 weeks)
* have dementia in accordance with DSM-V
* have either sleep/circadian rhythm disturbances, BPSD as identified by NPI-NH, or severely reduced ADL function
* provide written informed consent if the participant has capacity, if not, a written proxy informed consent from a legally authorized representative

Exclusion Criteria:

* are blind or may otherwise not benefit from light
* partake in another trial
* have a condition contra-indicated to the intervention
* have an advanced, severe medical disease/disorder and/or expected survival of less than 6 months or other aspects that could interfere with participation
* are psychotic or have a severe mental disorder

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-04-21 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Change in actigraphy recorded sleep and circadian rhythm | Baseline and week 8, 16, and 24
  An actigraph (Actiwatch 2, Philips Respironics) is worn for 7 consecutive days
Change in proxy-rated sleep | Baseline and week 8, 16, and 24
  Sleep Disorders Inventory (a proxy-rated instrument) is completed. A total score is calculated from the product of the average frequency and average severity of seven symptoms. The total score ranges from 0 (best) to 12 (worst).
Change in circadian rhythm of core body temperature | Baseline and week 8, 16, and 24
  A swallowed capsule (e-Celsius, BodyCap) records core body temperature for 24 hours.

SECONDARY OUTCOMES:
Change in the Neuropsychiatric Inventory - Nursing Home version (NPI-NH) | Baseline and week 8, 16 and 24
  NPI-NH is a proxy-rated instrument to assess neuropsychiatric disturbances in people with dementia. A total score is calculated from the product of the frequency and severity of 12 items. The total score ranges from 0 (best) to 144 (worst).
Change in the Cohen-Mansfield Agitation Inventory (CMAI) | Baseline and week 8, 16 and 24
  CMAI is a proxy-rated instrument measuring agitation symptoms. The instrument has 29 items, and the total score ranges from 29 (best) to 203 (worst).
Change in the Cornell Scale of Depression in Dementia (CSDD) | Baseline and week 8, 16 and 24
  CSDD is a proxy-rated instrument addressing depression in people with dementia. The instrument has 19 items, and the total score ranges from 0 (best) to 38 (worst).
Change in the Quality of Life in Late-Stage Dementia (QUALID) | Baseline and week 8, 16 and 24
  QUALID is a proxy-rated instrument validated for use in people with dementia. 11 behaviours are rated on a 5-point Likert scale, and the total score ranges from 11 (best) to 55 (worst).
Change in the Mobilization-Observation-Behaviour-Intensity-Dementia 2 (MOBID-2) | Baseline and week 16 and 24
  MOBID-2 is a proxy-rated instrument to assess pain in people with dementia. The instrument consists of two parts, each with five items. In part 1, pain intensity is inferred by the patient's pain behaviours during standardized, guided movements. In part 2, pain intensity is assessed by the patient's pain behaviours related to internal organs, head, and skin. A total score, ranging from 0-10, is set based on an overall assessment of the pain intensity scores in part 1 and 2.
Change in the Mini Mental State Examination (MMSE) | Baseline and week 24
  MMSE is a cognitive function screening instrument, which discerns severity of cognitive impairment on a 30 point scale. Lower scores represent severe impairment.
Change in the Functional Assessment Staging (FAST) | Baseline and week 8, 16 and 24.
  FAST is a proxy-rated instrument validated for use in people with dementia. It ascertains the severity of dementia in seven stages of functioning.
Change in the Physical Self-Maintenance Scale | Baseline and week 8, 16 and 24
  Physical Self-Maintenance Scale assesses Activities of Daily living (ADL) pertaining to physical function. The scale consists of six items, and the total score ranges from 0 to 30. Lower values indicate better functioning.
Clinical Global Impression of Change (CGIC) | Week 8, 16 and 24
  Rates globally perceived improvement ranging from very much worse (0) to very much improved (6). From baseline to week 8, 16 and 24.
Change in the Resource Utilization in Dementia - Formal Care (RUD-FOCA) | Baseline and week 8, 16 and 24
  RUD-FOCA is a cost-analysis of time invested in care during 24 hours
Change in general health | Baseline and week 8, 16 and 24
  The medical journal will be used to register change in total use of medication, blood pressure, pulse, weight and diagnoses.
Change in burden of care | Baseline and week 8, 16 and 24
  The NPI-NH total disruptiveness score is calculated by adding the occupational disruptiveness scores for the 12 items of the NPI-NH (each scored 0-5). The total disruptiveness score has a range of 0-60, with higher values representing more occupational disruptiveness.
Change in staff alertness | Baseline and week 8, 16 and 24
  Karolinska Sleepiness Scale comprises a single item assessing state sleepiness on a scale from 1 (very alert) to 9 (very sleepy, fighting sleep).
Change in staff sleep | Baseline and week 8, 16 and 24
  Bergen Insomnia Scale consists of six items. Each item is scored from 0 to 7, according to the number of days per week a specific insomnia symptom has occurred during the last month. The total score ranges from 0-42.
Change in staff fatigue | Baseline and week 8, 16 and 24
  The Chalder Fatigue Questionnaire has 13 items. The first 11 items (scored 0-3) are used to calculate a total score with a range from 0-33. Higher values represent more fatigue.
Change in staff mental health | Baseline and week 8, 16 and 24
  Measured by Hospital Anxiety and Depression Scale (HADS). HADS consists of two subscales, one for anxiety and one for depression, each with 7 items. The subscale scores range from 0 to 21. Higher values represent worse mental health (anxiety/depression).
Change in staff health related quality of life | Baseline and week 8, 16 and 24
  The SF-12 health survey consists of 12 items. Two summary scores (the Mental Health Component Summary and the Physical Health Component Summary) are calculated based on an algorithm from the User's Manual for the SF-12 Health Survey.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Flo, PhD, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Hordaland, Norway

REFERENCES:
- [Derived] Kolberg E, Hjetland GJ, Thun E, Pallesen S, Nordhus IH, Husebo BS, Flo-Groeneboom E. The effects of bright light treatment on affective symptoms in people with dementia: a 24-week cluster randomized controlled trial. BMC Psychiatry. 2021 Jul 28;21(1):377. doi: 10.1186/s12888-021-03376-y. PMID 34320937
- [Derived] Hjetland GJ, Kolberg E, Pallesen S, Thun E, Nordhus IH, Bjorvatn B, Flo-Groeneboom E. Ambient bright light treatment improved proxy-rated sleep but not sleep measured by actigraphy in nursing home patients with dementia: a placebo-controlled randomised trial. BMC Geriatr. 2021 May 17;21(1):312. doi: 10.1186/s12877-021-02236-4. PMID 34001024
- [Derived] Hjetland GJ, Nordhus IH, Pallesen S, Cummings J, Tractenberg RE, Thun E, Kolberg E, Flo E. An Actigraphy-Based Validation Study of the Sleep Disorder Inventory in the Nursing Home. Front Psychiatry. 2020 Mar 13;11:173. doi: 10.3389/fpsyt.2020.00173. eCollection 2020. PMID 32231600